CLINICAL TRIAL: NCT07072065
Title: Impact of Intralesional Tuberculin PPD Injection on Anogenital Warts: Interferon-Α, Interleukin-2, And Treatment Outcomes
Brief Title: Impact Of Intralesional Tuberculin Ppd Injection On Anogenital
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DV-202506.02
Record Dates: First submitted 2025-06-20; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Human Papilloma Virus; Infections
MeSH Terms: conditions — Infections | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGW patient treated with PPD antigen injection (Experimental): The PPD group received intralesional TPPD therapy, administering 5 TU (0,25 ml of PPD-2TU) to the largest AGW lesion once a week for six consecutive injections.
  Interventions: Drug: protein purified derivative
- AGW patient (No Intervention): Lesion observation for 6 week

INTERVENTIONS:
Drug: protein purified derivative — tuberculin purified protein derivative with dose 5 tuberculin unit
  Arms: AGW patient treated with PPD antigen injection

SUMMARY:
This clinical study investigates the immunological effects of tuberculin purified protein derivative (TPPD) therapy in patients with anogenital warts (AGW) caused by human papillomavirus (HPV).

Twelve AGW patients received intralesional TPPD injections (5 tuberculin units) once weekly for six weeks and were compared with twelve control patients.

Tissue samples were collected at baseline and after two injections for immunohistochemical analysis of interferon-alpha (IFN-α) and interleukin-2 (IL-2) expression.

Blood samples were collected at baseline and after six injections to measure serum levels of IFN-α and IL-2 using ELISA.

The study aims to evaluate TPPD as a potential immunotherapeutic agent by assessing cytokine responses associated with AGW regression.

DETAILED DESCRIPTION:
The research was conducted, in the STIs clinic at the Department of Dermatology and Venereology, Dr. Hasan Sadikin Hospital Bandung. The specimen was taken from 12 patients with AGW who have been previously treated with TPPD intralesional therapy, and 12 patients with AGW which not treated with TPPD as a control, from previous research titled which has received ethical clearance from Dr. Hasan Sadikin Hospital Bandung No. LB.02.01/X.6.5/291/2019.

The research inclusion criteria include specimen taken from patient with HPV infection in the anogenital area who have previously demonstrated a response to a 2 TU (0.1 ml) intradermal PPD antigen injection on the left forearm, with a minimum induration of 5 mm observed within 48-72 hours, and patients who were 12 years of age or older. Exclusion criteria include specimen from patient with a history of severe hypersensitivity reactions, such as anaphylaxis, to PPD antigen; pregnant or breastfeeding women; or who have received any other AGW treatments in the two to three months prior; those with immunosuppressive conditions or those who are taking immunosuppressive medications; patients with a history of asthma or other allergic conditions, as well as those experiencing active infections or other systemic illnesses; and patients with a history of keloids or seizures. The PPD group received intralesional TPPD therapy, administering 5 TU (0,25 ml of PPD-2TU) to the largest AGW lesion once a week for six consecutive injections. The technique involved positioning the syringe needle parallel to the skin surface, with the bevel facing upward. Evaluation of IFN-α and IL-2 expression was performed on AGW tissue and serum samples from AGW patients in the TPPD-treated group, both before and after therapy. Tissue cytokine expression was assessed after the second injection (week 2), while serum cytokine levels were measured after the sixth injection (week 6)

ELIGIBILITY:
Inclusion Criteria:

* Patients with HPV infection in the anogenital area.
* Prior positive response to a 2 TU (0.1 mL) intradermal PPD antigen injection on the left forearm, indicated by a minimum induration of 5 mm within 48-72 hours.
* Age 12 years or older.

Exclusion Criteria:

* History of severe hypersensitivity reactions (e.g., anaphylaxis) to PPD antigen.
* Pregnant or breastfeeding women.
* Received any other AGW treatments within the past 2-3 months.
* Immunosuppressive conditions or currently taking immunosuppressive medications.
* History of asthma or other allergic conditions.
* Presence of active infections or other systemic illnesses.
* History of keloids or seizures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Tissue IFN-α Expression in AGW Lesions (Measured by IHC) | Baseline and Week 2
  Quantification of IFN-α positive lymphocytes in anogenital wart (AGW) tissue samples using immunohistochemistry. The average number of IFN-α positive cells will be calculated from three high-power fields (400× magnification).
Change in Tissue IL-2 Expression in AGW Lesions (Measured by IHC) | Baseline and Week 2
  Quantification of IL-2 positive lymphocytes in AGW tissue samples using immunohistochemistry. Results are expressed as the mean number of positive cells across three high-power fields
Percentage Reduction in AGW Lesion Volume | Baseline to Week 6
  Lesion volume reduction calculated using the formula:
  [(Baseline Volume - Volume at Week 6) / Baseline Volume] × 100%.
  Therapeutic response will be classified as:
  No response: 0% reduction
  Minimal response: <50% reduction
  Partial response: 50-99% reduction
  Complete response: 100% reduction
Change in Serum IFN-α Levels (Measured by ELISA) | Baseline and Week 6
  Concentration of IFN-α in serum samples measured using a quantitative sandwich ELISA. Results will be reported in pg/mL.
Change in Serum IL-2 Levels (Measured by ELISA) | Baseline and Week 6
  Concentration of IL-2 in serum samples measured using a quantitative sandwich ELISA. Results will be reported in pg/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Venereology Clinic, Dr. Hasan Sadikin Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No